CLINICAL TRIAL: NCT07387575
Title: Screening for Intracranial Unruptured Aneurysms in First-Degree Relatives of Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Screening in Relatives With Elevated Risk for Unruptured Intracranial Aneurysms
Acronym: SIREN
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Novi Sad (Other)
Collaborators: Clinical Center of Vojvodina (Other)
Responsible Party: Principal Investigator, Nebojsa Lasica, Medical Doctor, University of Novi Sad
Other Study IDs: 00-18
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysms; Subarachnoid Hemorrhage, Aneurysmal
Keywords: Stroke; Intracranial Aneurysm; Brain Aneurysm; Familial Intracranial Aneurysm; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: 150 individuals that are first-degree relatives of affected patients admitted to study center for aneurysmal stroke and 150 individuals with sporadic UIAs

SUMMARY:
The purpose of this study is to screen first-degree relatives of patients with aneurysmal subarachnoid hemorrhage using magnetic resonance angiography to detect unruptured intracranial aneurysms. This study aims to identify individuals who are at increased risk and determine the effect of environmental factors for development of unruptured intracranial aneurysms.

DETAILED DESCRIPTION:
The prevalence of intracranial aneurysms is 3-5% according to studies, while the annual incidence of complications in the form of bleeding from an intracranial aneurysm is 8-10 per 100 000 people. Subarachnoid hemorrhage is an urgent condition characterized by the extravasation of blood into the space surrounding the central nervous system, which is filled with cerebrospinal fluid. The leading cause of non-traumatic subarachnoid hemorrhage is the rupture of an intracranial aneurysm, accounting for approximately 80-85% of cases, and it is associated with a high rate of complications and mortality. Therefore, early detection of patients at elevated risk, monitoring, and management of unruptured intracranial aneurysms is of paramount importance.

Data suggest that first-degree relatives of a family member affected have higher risk for developing intracranial aneurysm. Screening in Relatives with Elevated Risk for Unruptured Intracranial Aneurysms is research effort of neurosurgeons and neuroradiologists to identify environmental factors in study population of Vojvodina (Serbia), that contribute to development of intracranial aneurysms. This study will involve at least 150 siblings (first-degree relatives) of patients who suffered aneurysmal stroke, and determine effect of demographics, environmental factors including, smoking, medical comorbidities and hypertension, caffeinated drink consumption, and hard physical work on the development of unruptured intracranial aneurysms (UIAs). This study of affected families and individuals, known as Screening in Relatives with Elevated Risk for Unruptured Intracranial Aneurysms (SIREN) study, is sponsored by Provincial Secretariat of Health of the Autonomous Province of Vojvodina (Special Screening Program).

This study will also involve at least 150 individuals with no past family history of aneurysmal stroke or UIAs. SIREN study will take part in Autonomous Province in Vojvodina only.

In order to be eligible for the study, individuals with affected family member that was admitted to study center for aneurysmal stroke, had to be older than 30 years of age, and first-degree relatives (father, mother, sister, brother, daughter, or son).

Participants will be asked to complete informed consent and questionnaire with past medical and family history. After completing questionnaires, their arterial blood pressure will be measured. Participants will receive no monetary compensation for participation.

Identification of demographic and environmental risk factors contributing to development of UIAs in families of affected individuals may result in early detection of ones at risk and potentially prevent formation of UIAs or complications including aneurysmal stroke.

ELIGIBILITY:
Inclusion Criteria:

1. First-degree relatives (parents, siblings, or children) of patients diagnosed with aneurysmal subarachnoid hemorrhage (aSAH);
2. Age ≥ 30 years at the time of enrollment, and current cigarette smokers or diagnosed with hypertension (either treated or untreated);
3. Able and willing to undergo magnetic resonance angiography (MRA);

5. Able to provide written informed consent; 6. Sporadic aneurysm subjects must have a confirmed UIAs

Exclusion Criteria:

1. History of intracranial aneurysm rupture or prior subarachnoid hemorrhage;
2. Contraindications to MRI/MRA (e.g., pacemaker, metallic implants, severe claustrophobia) or pregnancy (due to MRI safety considerations);
3. A history of polycystic kidney disease, Marfan's Syndrome, Ehlers Danlos Syndrome, or fibromuscular dysplasia;
4. Unable or unwilling to provide informed consent;
5. Participation in another interventional study that could interfere with outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll first-degree relatives of patients with aneurysmal stroke who are aged 30 years or older, current smokers or have hypertension and individuals with sporadic UIAs and no past family history of aneurysmal stroke or UIAs. Participants must be able to undergo magnetic resonance angiography (MRA) and provide informed consent. Individuals with a prior intracranial aneurysm rupture, contraindications to MRI/MRA, pregnancy, or history of polycystic kidney disease, Marfan's Syndrome, Ehlers Danlos Syndrome, or fibromuscular dysplasia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Detection of unruptured intracranial aneurysms by magnetic resonance angiography (MRA). | At the time of screening (single MRA examination)
  The proportion of screened first-degree relatives (aged ≥30) who are found to have one or more UIAs.

SECONDARY OUTCOMES:
Correlation of aneurysm presence with risk factors | At the time of screening
  Analysis of the association between demographic and environmental (e.g., age, ethnicity, cigarette smoking, hypertension, consumption of caffeinated drinks, etc.) and the presence of UIAs.
Aneurysm size and location | At the time of screening
  Characterization of detected aneurysms by maximal size (millimeters) and anatomical location within the cerebral vasculature.
Prevalence of multiple aneurysms | At the time of screening
  Proportion of participants with multiple intracranial aneurysms (MIAs) detected on MRA. MIAs are defined as more than one UIAs in one patient.
Assessment of anatomical variations of cerebral arteries | At the time of screening
  Identification and classification of anatomical variations (e.g., vessel hypoplasia, fenestrations, duplicated arteries, circle of Willis variations, etc.) and evaluation of their association with the presence of UIAs.

CONTACTS AND LOCATIONS:
Overall Officials: Nebojsa M Lasica, M.D., Principal Investigator — University of Novi Sad
Locations (1):
- University Clinical Center of Vojvodina, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No